CLINICAL TRIAL: NCT06851182
Title: Comparison of Two Different Skin Stimulation Techniques on Intramuscular Injection Pain and Emotional Responses in Children: Helfer Skin Tap Technique and ShotBlocker
Brief Title: The Impact of Helfer Skin Tap and ShotBlocker Techniques on Emotional Responses to Intramuscular Injections in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, seher ÇEVİK, Assistant Professor, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Seher C Aktura
Record Dates: First submitted 2025-02-23; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Children
Keywords: Intramuscular Injection Pain; Emotional Responses in Children; Helfer Skin Tap Technique; ShotBlocker

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Helfer Skin Tap Group (Experimental): Helfer Skin Tap Group: The patient will be positioned in the most comfortable way possible. For the injection in the Vastus Lateralis muscle, the patient will be positioned appropriately lying down. After identifying the injection site, the skin will be gently tapped with the palmar surface of the dominant hand's fingers for approximately 5 seconds (about 15 strokes) to relax the muscles. After cleaning the skin with alcohol, the cap of the syringe in the dominant hand will be removed. The non-dominant hand's thumb and index finger will form a large V, and gentle taps will be applied to the skin again. The entire palm of the hand will be used to deliver three firm strokes to the muscle. The strokes (not slaps) should be firm to stimulate the large muscle fibers. After counting to three, the syringe will be inserted into the muscle at a 90° angle simultaneously.
  Interventions: Other: Helfer skin tap technique
- Shotblocker Group (Experimental): 1. Ensure that the patient takes the most comfortable position possible. For injection into the Vastus Lateralis muscle, the patient will be made to lie in the appropriate position.
  2. While removing the cap of the injector needle and holding it between the index and thumb of the active hand, the Shotblocker will be placed appropriately on the injection site with the passive hand, light pressure will be applied.
  3. The syringe will be inserted into the tissue smoothly at an angle of 90°. The needle will be prevented from moving in the tissue by holding the ajutage with the thumb and index finger of the passive hand. While holding the Shotblocker with the passive hand, the needle will be prevented from moving in the tissue by holding the ajutage with the thumb and index finger of the passive hand. Aspiration will be performed by pulling the piston back with the active hand.
  4. The drug will be injected into the muscle at a rate of 1ml/10sec.
  Interventions: Other: Shotblocker technique
- control (No Intervention): Children included in the control group will be administered IM Zofer drug (the drug will be injected into the muscle at a rate of 1ml/10 sec) with routine standard care of the ward.

INTERVENTIONS:
Other: Helfer skin tap technique — In the unit where the study was conducted, IM drug administration is performed through the Vastus Lateralis muscle in children aged 7-12 years and with BMI in the appropriate percentile according to age. No anaesthetic etc. application is performed. In order to create similar conditions in the study, children who are requested to be administered IM (ZOFER® 8mg / 4ml Injectable Solution-Ondansetron hydrochloride dihydrate into the Vastus Lateralis) will be included in the study. IM injection will be performed by the same investigator into the Vastus Lateralis muscle of the patient. A 16mm or 22mm, 22-25gauge sterile disposable sterile disposable needle will be used in all patients for injection administration. the procedure will be performed with helfer skin tap technique. Forms will be applied to the children by the researcher before and after IM injection.
  Other Names: Helfer skin tap
  Arms: Helfer Skin Tap Group
Other: Shotblocker technique — In the unit where the study was conducted, IM drug administration is performed through the Vastus Lateralis muscle in children aged 7-12 years and with BMI in the appropriate percentile according to age. No anaesthetic etc. application is performed. In order to create similar conditions in the study, children who are requested to be administered IM (ZOFER® 8mg / 4ml Injectable Solution-Ondansetron hydrochloride dihydrate into the Vastus Lateralis) will be included in the study. IM injection will be performed by the same investigator into the Vastus Lateralis muscle of the patient. A 16mm or 22mm, 22-25Gauge sterile disposable sterile disposable needle will be used in all patients. The procedure will be performed using Shotblocker method. Forms will be applied to the children by the investigator before and after IM injection.
  Other Names: Shotblocker
  Arms: Shotblocker Group

SUMMARY:
Study Aim: This study aims to determine the effects of the Helfer Skin Tap Technique (HST) and ShotBlocker application on pain, emotional indicators, and physiological parameters during intramuscular (IM) drug administration in children aged 7-12 years.

Study Design This research is designed as a randomized controlled experimental study.

Study Setting and Characteristics The study will be conducted at the Pediatric Emergency Clinic of Fırat University Hospital. The Pediatric Emergency Clinic consists of two observation rooms with a total of 12 beds, where children's medication administration and follow-ups are carried out.

The study population comprises children aged 7-12 years who received Vastus Lateralis IM drug administration (ZOFER® 8mg/4ml Injectable Solution - Ondansetron Hydrochloride Dihydrate) at the Pediatric Emergency Clinic of Fırat University Hospital and met the inclusion criteria during the specified study period.

For sample size estimation, the pain scores from the study by Sivri, Bilgen, and Balcı (2019) were considered. Based on their findings (d = 0.82; α = 0.05), it was determined that a sample size of 40 children per group (HST, ShotBlocker, and control) would be sufficient. Considering potential dropouts, the sample size was increased by 10%, and the study was planned to include a total of 132 children who met the inclusion criteria and provided informed consent along with their parents.

DETAILED DESCRIPTION:
This randomized controlled experimental study aimed to examine the effects of the Helfer Skin Tap Technique (HST) and ShotBlocker application on pain, emotional responses, and physiological parameters in children aged 7-12 years undergoing intramuscular (IM) drug administration. The study was conducted at the Pediatric Emergency Clinic of Fırat University Hospital between October 1, 2024, and January 31, 2025. The clinic consisted of two observation rooms with 12 beds, where children's medication administration and follow-ups were carried out. The study population included children aged 7-12 years who received Vastus Lateralis IM drug administration (ZOFER® 8mg/4ml Injectable Solution - Ondansetron Hydrochloride Dihydrate) and met the inclusion criteria.

The sample size was determined based on the pain scores from the study by Sivri, Bilgen, and Balcı (2019), with an effect size of d = 0.82 and α = 0.05, indicating that a sample of 40 children per group (HST, ShotBlocker, and control) was sufficient. To account for potential dropouts, the sample size was increased by 10%, resulting in a total of 132 children who met the inclusion criteria and provided informed consent along with their parents.

Participants' pre-test data were collected by the researcher before randomization. To ensure homogeneity, children were stratified based on age, gender, quality of life, and fatigue levels before being assigned to groups using a simple random sampling method. Blinding among researchers was not feasible, and patients in different groups were assigned to different hospital beds. To minimize selection bias, simple randomization was applied. The study protocol was registered in the ClinicalTrials.gov database, supported by the U.S. National Library of Medicine and the National Institutes of Health (NIH). Patients were unaware of their assigned groups (experimental or control).

Data Collection and Measurement Tools

Data were collected using the following tools:

Descriptive Characteristics Form (including age, gender, diagnosis, and history of IM injections).

Physiological Parameters Observation Form, which recorded pre- and post-injection heart rate, respiratory rate, and oxygen saturation using a pulse oximeter.

Faces Pain Scale-Revised (FPS-R), developed by Hicks et al. (2001), a self-reported scale ranging from 0 to 10, with higher scores indicating more severe pain.

Children's Emotional Indicator Scale (CEIS), developed by Li & Lopez (2005), measuring observable emotional behaviors in five categories (facial expression, vocalization, activity, interaction, and cooperation level), with scores ranging from 5 to 25, where higher scores indicated increased distress. The scale had a Cronbach's alpha value of 0.92 in its original version, while its Turkish adaptation in this study achieved 0.94.

Study Implementation IM injections were administered to children aged 7-12 years with a BMI percentile appropriate for their age. The injections were performed on the Vastus Lateralis muscle using a 16mm or 22mm, 22-25 gauge single-use sterile needle by the same researcher under standard conditions. No local anesthetic or analgesic was applied before the procedure. The research forms were completed before and after the injection by the researcher.

This study provided valuable insights into the effects of skin stimulation techniques on pain perception, emotional distress, and physiological responses in pediatric IM injections, contributing to improved pain management strategies in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* - 7 to 12 years old,
* BMI level in the appropriate range according to age,
* IM drug administered to the Vastus Lateralis muscle,
* No disease that causes chronic pain,
* Not taking any analgesic medication in the last 8 hours before the procedure,
* No mental or neurological disability,
* No visual or auditory problems preventing the application of the scales,
* Speaks and understands Turkish,
* Children whose parents and themselves agreed to participate in the study were included in the study.

Exclusion Criteria:

* - BMI level is not in the appropriate range according to age,
* Forms with incomplete or incorrect answers,
* Children who did not volunteer to participate in the study were excluded from the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Children's Emotional Indicator Scale | 1 month
  The Children's Emotional Indicator Scale (CEIS) was developed by Li and Lopez (2005) to provide a simple, objective and consistent method for nurses to identify children's emotional behaviors during stressful medical procedures. The CSA consists of five categories of observable emotional behaviors (Facial expression, Vocalization, Activity, Interaction and Level of cooperation). Each category has a value between 1-5. The total score that can be obtained from the scale varies between 5-25. The higher the scores obtained from the scale, the higher the negative emotional indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Cevik Aktura, Principal Investigator — Inonu University
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No